CLINICAL TRIAL: NCT01962922
Title: Prospective, Rand, Open-label, Single-center, 2 Sequence, 3 Period Crossover Study to Compare the Steady State PK of Once-Daily-Extended Release LCP-Tacro to Generic Tacrolimus Capsules Twice Daily in Stable A A Renal Transplant pt.
Brief Title: Crossover Study to Compare PK of Once Daily LCP-Tacro Tablets to Generic Tacrolimus Capsules Twice Daily.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Veloxis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LCP-Tacro 3004
Record Dates: First submitted 2013-10-08; First posted 2013-10-14 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LCP-Tacro (Active Comparator): Envarsus XR
  Interventions: Drug: LCP-Tacro
- Tacrolimus - IR (Active Comparator): Tacrolimus
  Interventions: Drug: Tacrolimus -IR

INTERVENTIONS:
Drug: LCP-Tacro — once-daily extended release tablet
  Other Names: Envarsus XR
  Arms: LCP-Tacro
Drug: Tacrolimus -IR — twice daily capsules
  Other Names: Prograf; Generic Tacrolimus
  Arms: Tacrolimus - IR

SUMMARY:
Open label, prospective, single-center, randomized, two sequence, three period crossover study to compare the steady state pharmacokinetics of LCP-Tacro tables to generic tacrolimus capsules administered twice daily in stable African-American renal transplant patients.

DETAILED DESCRIPTION:
This is open label, prospective, single-center, randomized, two sequence, three period crossover study to compare the steady state pharmacokinetics of once daily dosing of LCP-Tacro tablets to tacrolimus capsules administered twice daily in stable African American kidney transplant patients.

Approximately 72 male and female African American renal transplant patients on table immunosuppression regimens will be randomly assigned in a 1:1 ratio to one of two sequences:

Sequence 1: (n=36) 18 patients requiring less than 0.15 mg/kg/day and 18 patients requiring equal to or greater than 0.15 mg/kg/day. Patients will continue on generic tacrolimus capsules on days 1-7 (24 hours PK profile on day 7) then patients are switched to LCP-Tacro tablets (at 15% lower dose of twice daily generic tacrolimus) on day 8.

Sequence 2: (n=36) 18 patients requiring less than 0.15 mg/kg/day and 18 patients requiring equal to or greater than 0.15 mg/kg/day. Patients will receive LCP-Tacro tablets (at 15% lower dose than generic tacrolimus twice daily formulation) on days 1-7 (24 hour PK profile on day 7) patients are switched back to twice daily generic tacrolimus treatment beginning on day 8.

ELIGIBILITY:
Inclusion criteria:

* Age ≥18-80 old, male or female
* African Americans
* Willing to give written informed consent and to comply with study visits and restrictions, including being able to speak, write and understand English
* Pt who have received a primary or secondary transplant
* Pt least 6 (six) mth post-transplant and on a stable dose of tacrolimus
* BMI ≥19
* Pt who are sero-positive for Hepatitis B or C positive may also be enrolled
* Pt maintained on concurrent immunosuppression with stable doses during screening
* Pt on a proton PPI remain on the same PPI formulation and dose during the PK portion of the study.
* During PK phase Only: Pt taking any medication that could interfere with tacrolimus blood levels, including prescription and over-the-counter medications, herbal or food supplements (including grapefruit, and pomegranate products), or medications must continue the same dose and are willing to continue the same dose/routine
* During PK phase Only: the patient is not scheduled to begin any new medication that could interfere with tacrolimus blood levels, including prescription and over-the-counter medications, herbal or food

Exclusion Criteria:

* Evidence of acute rejection episode within the past three months
* Pt not Africa-American
* Recipients of organ transplants other than kidney
* Known to be HIV positive at transplant
* Pt with recurrent focal segmental glomerulosclerosis (FSGS)
* Pt with any severe medical condition (including infection) requiring acute or chronic treatment
* Pt with a positive DSA
* Pt with a positive BK virus results
* GFR < 25 ml/min measured by MDRD4 as SOC within last 30 days
* Patients with AST, ALT, total bilirubin > 2.5 x ULN or evidence of severe liver disease
* Pt with WBC < to 2000/mm3 or ANC < to 1500 mm3 with PLT < 75,000/mm3 or HGB < 8 g/dl
* Pt with mental or physical conditions or known non-adherence
* Presence of intractable immunosuppressant complications of side effects resulting in dose adjustment of tacrolimus
* Exposed to investigational therapy within 30 days prior to enrollment
* No anticipated changes in the immunosuppressive regimen, other than those specified by the study protocol
* Pt with severe diabetic gastroparesis or other severe GI disturbances
* Pt who have underwent gastric banding or gastric bypass at any time pre or post-transplant
* Pregnant or nursing (lactating) women, or planning to become pregnant
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant who are unwilling to use a defined SOC of method

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-11; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Callahan, RN, Study Director — Veloxis Pharmaceuticals
Locations (3):
- United States (3):
  - University of Illinois, Chicago, Chicago, Illinois
  - Washingto University School of Medicine, St Louis, Missouri
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trofe-Clark J, Brennan DC, West-Thielke P, Milone MC, Lim MA, Neubauer R, Nigro V, Bloom RD. Results of ASERTAA, a Randomized Prospective Crossover Pharmacogenetic Study of Immediate-Release Versus Extended-Release Tacrolimus in African American Kidney Transplant Recipients. Am J Kidney Dis. 2018 Mar;71(3):315-326. doi: 10.1053/j.ajkd.2017.07.018. Epub 2017 Nov 20. PMID 29162334

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 25 November 2013 (first patient enrolled) to 09-Mar-2015 (last patient completed initial pharmacokinetics [PK] portion of the study, the 'PK Cross-over' period), approximately 16 months enrolled from 3 US medical centers:University of Pennsylvania;University of Illinois at Chicago;Washington School of Medicine
Groups:
- Sequence 1: •Sequence I: (n=27) Patients will continue on twice-daily IR-Tac capsules on Days 1-7 (24-hour PK profile on Day 7), then patients are switched to Envarsus XR tablets (at a dose 15% lower than their Tac - IR doses) on Day 8. PK on day 14 and 21.
  Patients in sequence 1 are on Envarsus XR at Day 21. Patient may continue on extension up to a total of 6 months.
- Sequence 2: • Sequence II: (n=23) 1 Patients receive Envarsus XR tablets (at 15% lower dose than their IR-Tac dose) on Days 1-7 (24-hour PK profile on Day 7), then patients are switched back to twice-daily Tac - IR treatment beginning on Day 8. PK on days 14 and 21.
  Patients in sequence 2 are on Tac - IR at Day 21. Patient have option of continuing in extension portion of the study on Tac - IR for up to 6 months.
Period: PK Portion Day 7
Arm/Group | Sequence 1 | Sequence 2
Started | 27 | 23
Completed | 23 | 23
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — non-compliance | 1 | 0
Period: PK Portion Day 14
Arm/Group | Sequence 1 | Sequence 2
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0
Period: PK Portion Day 21
Arm/Group | Sequence 1 | Sequence 2
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0
Period: Extendion Portion (up to Month 6)
Arm/Group | Sequence 1 | Sequence 2
Started | 23 | 23
Completed | 18 | 20
Not Completed | 5 | 3
Not completed — no longer wished to participate in study | 4 | 3
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sequence I: Sequence I IR-Tac→Envarsus XR (N = 27)
- Sequence II: Sequence II Envarsus XR→IR-Tac (N = 23)
- Total: Total of all reporting groups
Arm/Group | Sequence I | Sequence II | Total
Number analyzed (Participants) | 27 | 23 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 20 | 46
  >=65 years | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 15 | 14 | 29
Region of Enrollment [Number; unit: participants]
  United States | 27 | 23 | 50

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of AUC(0-24) for Envarsus XR and IR-Tac
Description: Tacrolimus whole blood concentrations obtained from the central lab was used for PK analysis. Actual sampling time was used to calculate AUC(0-24). Arithmetic mean and standard deviation is given below.
  Nominal time points used were: Pre-dose (C0) and then 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 13, 14, 16, 18 and 24 hours.
Time Frame: Day 7
Population: For this outcome measure the PK population N=46 was used.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Envarsus XR: Tacrolimus tablets once daily.
- Tacrolimus - IR: Tacrolimus capsules twice daily.
Arm/Group | Envarsus XR | Tacrolimus - IR
Number analyzed (Participants) | 23 | 23
ng*hr/mL | 251.9 (77.78) | 247.9 (102.33)

2. Primary Outcome: Evaluation of C(Max) for Envarsus XR and IR-Tac
Description: Tacrolimus whole blood concentrations obtained from the central lab was used for PK analysis. Actual sampling time was used to calculate C(max). Arithmetic mean and standard deviation is given below.
  Nominal time points used were: Pre-dose (C0) and then 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 13, 14, 16, 18 and 24 hours.
Time Frame: Day 7
Population: For this outcome measuure the Protocol PK population of N = 46 was used.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Envarsus XR | Tacrolimus - IR
Number analyzed (Participants) | 23 | 23
ng/mL | 16.53 (5.464) | 26.84 (13.296)

3. Primary Outcome: Evaluation of C(Min) for Envarsus XR and IR-Tac
Description: as for outcome 1
Time Frame: Day 7
Population: For this outcome measure the Protocol PK population N= 46 was used.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Envarsus XR | Tacrolimus - IR
Number analyzed (Participants) | 23 | 23
ng/mL | 7.51 (2.487) | 7.06 (2.843)

4. Primary Outcome: Evaluation of AUC(0-24) for Envarsus XR and IR-Tac
Description: as for outcome 1
Time Frame: Day 14
Population: For this outcome measure the PK population N=46 was used
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Envarsus XR | Tacrolimus - IR
Number analyzed (Participants) | 23 | 23
ng*hr/mL | 293.3 (124.40) | 225.7 (56.27)

5. Primary Outcome: Evaluation of C(Max) for Envarsus XR and IR-Tac
Description: as for outcome 2
Time Frame: Day 14
Population: For this outcome measuure the Protocol PK population of N = 46 was used.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Envarsus XR | Tacrolimus - IR
Number analyzed (Participants) | 23 | 23
ng/mL | 20.83 (9.265) | 26.31 (13.296)

6. Primary Outcome: Evaluation of C(Min) for Envarsus XR and IR-Tac
Description: as for outcome 1
Time Frame: Day 14
Population: For this outcome measuure the Protocol PK population N= 46 was used.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Envarsus XR | Tacrolimus - IR
Number analyzed (Participants) | 23 | 23
ng/mL | 8.34 (3.769) | 6.46 (1.692)

7. Primary Outcome: Evaluation of AUC(0-24) for Envarsus XR and IR-Tac
Description: as for outcome 1
Time Frame: Day 21
Population: For this outcome measure the PK population N=46 was used.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Envarsus XR | Tacrolimus - IR
Number analyzed (Participants) | 23 | 23
ng*hr/mL | 289.3 (111.79) | 230.3 (53.83)

8. Primary Outcome: Evaluation of C(Max) for Envarsus XR and IR-Tac
Description: as for outcome 2
Time Frame: Day 21
Population: For this outcome measuure the Protocol PK population of N = 46 was used.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Envarsus XR | Tacrolimus - IR
Number analyzed (Participants) | 23 | 23
ng/mL | 19.71 (8.387) | 26.31 (7.871)

9. Primary Outcome: Evaluation of C(Min) for Envarsus XR and IR-Tac
Description: as for outcome 1
Time Frame: Day 21
Population: For this outcome measure the Protocol PK population N= 46 was used.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Envarsus XR | Tacrolimus - IR
Number analyzed (Participants) | 23 | 23
ng/mL | 8.01 (3.281) | 6.62 (1.692)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of first dose of study medication, through and including last dose of study medication during the up to 6 month extension period.
Description: Adverse events are associated with the treatment the patient is on at the onset date of the adverse event and not the portion of the study (e.g. PK or extention portion). The below figures are cumulative for the entire study participation start of study through 6 month extension.
Groups:
- Envarsus XR: Tacrolimus extended release
- Tacrolimus - IR: brand IR tacrolimus
Arm/Group | Envarsus XR | Tacrolimus - IR
Serious Adverse Events (participants affected / at risk) | 3/50 | 4/50
Other Adverse Events (participants affected / at risk) | 23/50 | 22/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Envarsus XR (N=50) | Tacrolimus - IR (N=50)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Otitis Media (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Envarsus XR (N=50) | Tacrolimus - IR (N=50)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Nasopharyngitis (Infections and infestations) | 3 (3) | 5 (5)
Blood creatinine increased (Investigations) | 7 (8) | 4 (4)
Glomerular filtration rate decreased (Investigations) | 5 (5) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 2 (3) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has no objection to publication of the results of the Study by Site based on information collected or generated by Site; provided, however, that such publication must not precede the primary manuscript (unless no such multi-site publication is completed within twelve (12) months following the completion of the Study or unless Sponsor notifies Site in writing that no such multi- center publication shall be made).